CLINICAL TRIAL: NCT02630381
Title: Treatment of Osteoporosis With Unfocused Extracorporeal Shock Wave Therapy: Pilot Study
Brief Title: Shock Wave Therapy for Osteoporosis
Acronym: BOEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Marianne Koolen, Drs, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL40580.078.12
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Osteoporosis
Keywords: high-energy shock waves
MeSH Terms: conditions — Osteoporosis | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Shock wave arm (Experimental): Unfocused extracorporeal shock wave therapy will be applied on the distal radius on one site when the patient is receiving general anaesthesia for surgery on the lower extremity or spine.
  Interventions: Device: Unfocused extracoporeal shock wave therapy
- Contra-lateral arm (No Intervention): The distal radius and/or wrist that did not receive UESWT will not be treated

INTERVENTIONS:
Device: Unfocused extracoporeal shock wave therapy — Shock waves are acoustical pulses that are characterized by high amplitude (~500 bar) and short rise time (~20 ns), which are followed by a longer low-magnitude negative wave (~-100 bar). Extracorporeal shock waves are widely used to disintegrate kidney stones, which is called lithotripsy. In orthopedics, shock wave therapy, called orthotripsy, is used safely in a variety of musculoskeletal disorders like non unions, osteonecrosis of the hip, Achilles and patellar tendinopathy, lateral epicondylitis of the elbow and fasciitis plantaris.
  Until recently extracorporeal shock wave therapy for musculoskeletal disorders was applied with a focused character, in which the waves converge in a focal point similar to lithotripsy. For the prevention of fractures in osteoporosis a focused character is not preferable because large skeletal regions have to be treated, so unfocused shock waves have been developed.
  Other Names: Extracorporeal shock waves; Extracorporeal shock wave therapy
  Arms: Shock wave arm

SUMMARY:
Rationale: Osteoporotic fractures are associated with high morbidity and mortality. This is why prevention of these fractures is important. The investigators have shown in animal studies that a single treatment with unfocused extracorporeal shock wave therapy leads to highly increased bone mass and improved biomechanical properties. Unfocused extracorporeal shock wave therapy could have important implications for the prevention of osteoporotic fractures.

Objective: To assess the effect of unfocused extracorporeal shock wave therapy on bone mass.

Study design: A clinical pilot study. Study population: Twelve female patients are eligible if they are undergoing elective surgery of the lower extremity or elective spinal surgery under general anesthesia in the investigators hospital.

Intervention: When the patient is under general anaesthesia he/she will receive 3000 unfocused extracorporeal shock waves (energy flux density 0.3mJ/mm2) to one distal forearm. The contra lateral forearm will not be treated and serves as a control.

Main study parameters/endpoints:

The investigators will examine the effect on bone mass with the use of repeated dual energy X-ray absorptiometry measurements. These results are necessary to calculate the number of patients that are needed for larger studies. Furthermore, the investigators will assess patient's discomfort.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: General anaesthesia is performed during treatment and pain after the procedure will be evaluated using pain scales and, if necessary pain medication will be prescribed by the orthopaedic surgeon. The dual energy X-ray absorptiometry-scans and X-rays will cause very low radiation exposure to the patient.

ELIGIBILITY:
Inclusion Criteria:

* female sex, age 50-80 years, normal dietary intake inclusive calcium and/or milk products and willing to participate

Exclusion Criteria:

* skin disease, systemic corticosteroid use, known systemic disease that interacts with bone (eg. rheumatoid arthritis, multiple myeloma, hyper(para)thyroidism, Paget's disease or Cushing's disease) or a previous wrist fracture

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
Bone mineral density will be assessed with the use of repeated dual energy X-ray absorptiometry measurements | 12 weeks
Bone mineral density will be assessed with the use of repeated dual energy X-ray | 6 weeks

SECONDARY OUTCOMES:
Pain on the VAS scale | day before and first week after treatment
Patient's side effects and complications on a questionnaire | 12 weeks